CLINICAL TRIAL: NCT03563261
Title: Interactions of Muscle-Tendon Mechanics During Stair Climbing and Trip Recovery, and Efficacy of Collagen Supplementation for Functional Improvement for Older Adults
Brief Title: Muscle-Tendon Mechanics During Locomotor Tasks, Efficacy of Collagen Supplementation for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Heloise Debelle, Principal Investigator, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Collagen_OA_V1
Record Dates: First submitted 2018-05-15; First posted 2018-06-20 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Tendon Stiffness With Age
Keywords: Older Adults; Collagen supplementation; Locomotor behaviour

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized control study
Who Masked: Participant, Investigator
Masking Description: Participants and researchers will not know if participants are allocated to the control or active product group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen supplement group (Active Comparator): Participants assigned in the collagen supplement group will drink the active product every morning before breakfast.
  Interventions: Dietary Supplement: Collagen supplement group
- Placebo supplement group (Placebo Comparator): Participants assigned in the placebo supplement group will drink the placebo every morning before breakfast.
  Interventions: Dietary Supplement: Placebo supplement group

INTERVENTIONS:
Dietary Supplement: Collagen supplement group — Participants from both group will take their supplement every morning prior to breakfast. Supplementation period will be 4 months. They will perform tendons loading activities 30 minutes after ingestion of the supplement. Tendons loading activities will be heel raises and knee extensions while seated. Participants will be asked to keep the exercise intensity low as it is not a strengthening intervention.
  Arms: Collagen supplement group
Dietary Supplement: Placebo supplement group — Participants from both group will take their supplement every morning prior to breakfast. Supplementation period will be 4 months. They will perform tendons loading activities 30 minutes after ingestion of the supplement. Tendons loading activities will be heel raises and knee extensions while seated. Participants will be asked to keep the exercise intensity low as it is not a strengthening intervention.
  Arms: Placebo supplement group

SUMMARY:
Older adults are at higher risks of tripping and falling than young adults. These falls may lead to serious injuries (bone fractures, head trauma…) and premature death. They also have an important economic cost for the society. One of the reasons identified for this increased risk of falling is the modification of muscles and tendons functional and architectural parameters with age. It is now well established that muscles of older adults are smaller and weaker, while tendons, that modulate the outcomes of muscle contraction, are less able to resist to tension and transmit forces more slowly than in young age. These changes have functional implications, especially in tasks that require to quickly generate high forces, such as recovering from a trip.

This study aims to determine the links between muscle-tendon characteristics and locomotion, and to understand whether they can be improved by a four-months collagen supplementation.

The investigators will measure the muscular strength and tendon stiffness of lower limb musculotendinous units (MTU) for older adults using isokinetic dynamometry (IKD) and ultrasounds. Participants' abilities to recover from a trip will then be evaluated using a custom built tripping device while walking on a treadmill (participants will wear a whole body harness attached to a rope secured to the ceiling). These performances will be linked to MTU characteristics and compared between both age groups. Finally, the investigators will evaluate the effect of a nutritional supplementation on the mechanical properties of elderly tendons and its potential impacts on their ability to safely recover from a trip, on their lean mass, and on other life quality related markers (joint pain, balance, stair climbing capacities...).

The investigators expect that this study will lead to a new intervention aiming to improve the safety of older adults performing their daily activities using nutritional supplementation, which is known to have better adherence than training interventions.

DETAILED DESCRIPTION:
Being able to walk safely, to go up and down stairs and to recover from an unexpected gait perturbation are vital for older adults' autonomy, home maintenance and life quality. It is therefore of major interest to understand the mechanisms responsible for older adults (OA) decreased functional abilities. This study aims first to understand the links between muscles and tendons characteristics and functional capacities of OA, and second to evaluate whether a 4-month collagen supplementation can improve OA musculotendinous properties, thereby improving their function.

Trips are caused by an unexpected perturbation during the swing phase of gait (i.e. when the foot is not in contact with the ground). Recovering from a trip requires the production of fast and large muscle torques at the hips, knees and ankles joints to counteract the forward rotation of the body, and the propulsion of the forward leg anteriorly to the centre of mass.

For OA, falling when walking on a flat surface is potentially damaging, and falling while using stairs is even more dangerous. Indeed, over 65% of falls leading to brain injury in OA happen in stairs and 10% of fall death in the US happen in stairs. Older adults with joints problem are more susceptible to report difficulties when using stairs than those without. Those with multiple joints problems are also up to 20 times more likely to have difficulties in stair climbing than OA without joint problems. Mechanically, older adults operate closer to their maximal joint moment capacities at the knee (ascent and descent) and ankle (ascent). They thus have less reserve to adjust to any perturbation that could happen and are at more risks of falling than young adults (YA).

Normal gait, but also trip recovery and stair climbing are dependent on the muscles and tendons capacities to produce and transmit adequate forces in a short amount of time.

With age, muscular and tendinous properties decline: muscles, that are responsible for the production of forces, become weaker and smaller, and tendons, that are responsible for the transmission of forces from muscles to the skeleton, become less stiff. It has been shown that changes in the gastrocnemius tendon's properties affect the ability of elderly to maintain balance during dynamic and demanding postural tasks, complicating OA daily living activities. This may especially be so when the individual is not only required to generate large joint moments, but to do so quickly, as is the case when trying to avoid a fall. OA with decreased muscle and tendon properties do not generate and transmit adequate forces in magnitude and velocity, which may be responsible for their decreased ability to recover from a trip and in some cases may lead to falls. Therefore, interventions that improve muscle-tendon properties of OA are likely to have benefits for recovering from a trip and preventing a fall occurring.

Training interventions have been developed to minimise the effect of age on OA physical condition but although strength training can improve tendon stiffness and muscle strength, participants' adherence to these protocols can be low. Developing interventions with similar effects and which are easier to follow (that do not require modification of participants' routine) is thus of major interest.

It has been shown that collagen supplementation improves the blood collagen synthesis and the resistance to tension of collagenous tissues in the body. In this study, the investigators will test a collagen supplement designed to improve joint, muscle and whole-body function.

Although the investigators understand that the structure of muscles and tendons determines their function and has key roles in overall physical function and ability to recover from a trip, the investigators do not yet fully understand these mechanisms and how best to improve them. The research area will be centred upon the muscle-tendon properties and interactions that determine physical function in two different conditions (stair climbing and trip recovery), and whether these can be improved by collagen supplementation.

The investigators will therefore evaluate changes in bone mineral density, lean mass, tendon stiffness, muscle strength, stair climbing and tripping recovery capacities before and after a 4-month supplementation period in 80 OA allocated either to the active product or to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 50 years
* Mean age: maximum 65 years

Exclusion Criteria:

* Any lower limb injury in the last 6 months
* A joint replacement
* Neural, musculoskeletal or balance disorder that could affect the musculoskeletal system or capacity to execute functional tasks
* Be taking any nutritional supplements that affect muscle or tendon size or function or stopped its intake less than 3 months before the baseline
* Presence of systemic diseases (e.g., diabetes mellitus or cardiovascular, kidney, liver or lung disease)
* Pregnant or breast feeding
* History of drug abuse
* Taking anti-inflammatory medication within 24 hours the baseline
* Allergic to any ingredient in the test products (meat, fish or soy)
* Concurrent participation in other clinical studies
* Taking medication to treat a chronic disease (e.g., rheumatoid arthritis, psoriatic arthritis, fibromyalgia, gout and inflammatory joint disease for example bursitis or tennis elbow, and any other type of chronic pain syndrome other than osteoarthritis)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Tendon stiffness | at baseline and after the end of the supplementation period (4-months)
  Tendon stiffness will be measured as the change in tendon length per change in tendon force. Tendon lengthening will be measured using B-mode ultrasound as the displacement of the proximal insertion (myotendinous junction (MTJ) for the Achilles tendon and patellar insertion for the patellar tendon) during maximum voluntary contractions.

SECONDARY OUTCOMES:
Rate of torque development (RTD) | at baseline and after the end of the supplementation period (4-months)
  RTD is dependant of tendon stiffness and is measured as the gradient of the torque-time curve during isometric contractions.
Muscles strength | at baseline and after the end of the supplementation period (4-months)
  Muscle strength will be measured during isometric and isokinetic (concentric) contractions and will be used to plot the force-velocity profile of each participant.
Muscle length | at baseline and after the end of the supplementation period (4-months)
  Muscle length will be measured at rest using B-mode ultrasounds images captured at the proximal and distal insertions. Muscle length will be measured as the straight line between these 2 points.
Fascicle length | at baseline and after the end of the supplementation period (4-months)
  Fascicle length will be measured using B-mode ultrasounds. Ultrasound images will be captured at the mid belly of the muscle. Fascicle length will be defined as the straight line distance between the upper and the lower aponeurosis parallel to the lines of collagenous tissue.
Muscle cross sectional area | at baseline and after the end of the supplementation period (4-months)
  Cross sectional area will be measured at rest using B-mode ultrasounds. Transversal-planed images will be captured.
Pennation angle | at baseline and after the end of the supplementation period (4-months)
  Pennation angle will be measured using B-mode ultrasounds. Ultrasound images will be captured at the mid belly of the muscle. Pennation angle will be defined at the angle between the fascicle and the lower aponeurosis.
Tendon length | at baseline and after the end of the supplementation period (4-months)
  Tendons length will be measured at rest using B-mode ultrasounds. Tendon length will be measured as the distance between the proximal and the distal ends.
Tendon cross sectional area | at baseline and after the end of the supplementation period (4-months)
  Cross sectional area will be measured at rest using B-mode ultrasounds. Tendon cross sectional area will be measured by transversal plane scanning at 25, 50 and 75% of tendon length.
EMG (Electromyography) activity | at baseline and after the end of the supplementation period (4-months)
  EMG activity will be measured during muscle contractions using electrodes placed on the skin. EMG activity represents the electric activity of a muscle.
Electromechanical delay | at baseline and after the end of the supplementation period (4-months)
  Electromechanical delay will be measured during muscle contractions using electrodes placed on the skin. The electromechanical delay (EMD) corresponds to the time latency between the beginning of muscle activation and the beginning of moment development, quantified by visual inspection of the EMG and force-time traces.
Whole body bone mineral density | at baseline and after the end of the supplementation period (4-months)
  Bone mineral density will be measured using DXA (Dual-energy X-ray absorptiometry) scan
Lean mass | at baseline and after the end of the supplementation period (4-months)
  Lean mass will be measured using the same DXA (Dual-energy X-ray absorptiometry) scan
Balance | at baseline and after the end of the supplementation period (4-months)
  Berg balance scale, which is a test aiming to evaluate balance among older people, will be used to evaluate objectively participants balance while performing different tasks (standing with eyes closed, standing on one foot, retrieving object from floor…). Each task is evaluated on 4 points: such as 4 points represent a good balance and 0 point a poor balance. Fourteen tasks have to be completed with a total score of 56. Participants ranging from 0 to 20 are considered as being at high risk of falling (poor balance), those ranging from 21 to 40 as being at medium risk of falling and those ranging from 41 to 56 as low risk of falling (good balance).
  Total score: Scores for each task will be summed to obtain the total score. MAXIMUM total score = 56.
Participants' confidence for activities-specific balance tasks | at baseline and after the end of the supplementation period (4-months)
  Participants' confidence for activities-specific balance tasks will be evaluated using the ABC-scale (activities specific balance confidence scale): they will have to rate their balance confidence for performing activities by answering to the question 'How confident are you that you will not lose your balance or become unsteady when you…' for several tasks such as walking around the house, walking up or down stairs… For each activity, participants will have to indicate their level of confidence in doing the activity without losing their balance or becoming unsteady from choosing one of the percentage points on the scale from 0% to 100% (0% represents no confidence and 100% represents complete confidence).
  Percentages obtain for each question (total 16 questions) will be summed and the total divided by 16 to obtain each subject's ABC score.
Knee scoring scale | at baseline and after the end of the supplementation period (4-months)
  Lysholm Knee Scoring Scale questionnaire will be used to evaluate how participants' knee problems have affected their ability to manage in everyday life. For each question they will have to choose the answer that best applies to them at the moment. The total score is the sum of each response to the questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability. Lower scores indicate a worse outcome with more symptoms or disability.
Joints pain | at baseline and after the end of the supplementation period (4-months)
  A numerical rating scale (NRS) will be used to evaluate participants' joints pain.
  They will first have to answer (Yes or No) to the question:
  Do you usually suffer from any joint pain?
  If the answer is YES, they will have to specify which joints are usually painful and where appropriate which side. Joints investigated are the following: shoulder, elbow, wrist, hand, back, lower back, neck, hip, knee, ankle and foot.
  For each painful joint (and each side), participants will have to rate from 0 to 100 the amount of pain they had in the last 24 hours. 0 being no pain at all and 100 the worst pain possible.
Participants' perceived risk of falling | at baseline and after the end of the supplementation period (4-months)
  The fall efficacy scale international (FES-I) will be used to measure participants' perceived risk of falling. Participants will have to answer to the question "How concerned are you about the possibility of falling when you are…?" for 16 items. For each item, the score goes from 1 to 4, 1 being not at all concerned, 2 being somewhat concerned, 3 being fairly concerned and 4 being very concerned. The sum of all scores gives a maximum total of 64 points. A higher score indicates a greater fear of falling.
Participants' health perception | at baseline and after the end of the supplementation period (4-months)
  The Nottingham Health Profile will be used to measure participants' health perception. It provides a brief indication of participants' perceived emotional, social and physical health problems. The questionnaire is composed of 38 questions for which participants have to answer "Yes" or "No" in 6 subareas (energy level, pain, sleep, social isolation, physical abilities and emotional reaction). A weighted value is assigned to each question. The sum of all weighted values in a given subarea adds up to 100. The higher the score, the greater the number and severity of problems.
Trip recovery: step length | at baseline and after the end of the supplementation period (4-months)
  Step length will be quantified from the kinematic data obtained during trip recovery
Trip recovery: margin of stability | at baseline and after the end of the supplementation period (4-months)
  Margin of stability during trip recovery will be measured using the centre of pressure displacement.
Trip recovery: number of steps required to be back to baseline | at baseline and after the end of the supplementation period (4-months)
  Number of steps required to be back to baseline margin of stability will be measured using a motion capture system.
Trip recovery: joint moments | at baseline and after the end of the supplementation period (4-months)
  Joint moments during trip recovery will be measured using kinematic and kinetic data obtained during the gait analysis
Trip recovery: joint power | at baseline and after the end of the supplementation period (4-months)
  Joint power during trip recovery will be measured using kinematic and kinetic data obtained during the gait analysis
Trip recovery: EMG activity | at baseline and after the end of the supplementation period (4-months)
  EMG activity of lower limb muscles (gastrocnemius, quadriceps, soleus, biceps femoris) will be measured using electrodes placed on the skin.
Trip recovery: MTJ displacement | at baseline and after the end of the supplementation period (4-months)
  Musculotendinous junction (MTJ) displacement will be measured during trip recovery using B-mode ultrasound images.
Stair climbing: centre of pressure to centre of mass distance | at baseline and after the end of the supplementation period (4-months)
  Centre of pressure to centre of mass distance during stair climbing will be measured from the kinematic data obtained during stair climbing.
Stair climbing: pain level | at baseline and after the end of the supplementation period (4-months)
  Participants' degree of pain while using the staircase will be evaluated using a numerical rating scale.
  They will first have to answer by Yes or No to the question:
  Now that you have used the staircase, did it trigger any joint pain? If yes, they will have to specify which joint was painful, and where appropriate which side. Joints investigated are the following: back, lower back, hip, knee, ankle and foot.
  For each painful joint (and each side), participants will have to rate from 0 to 100 their amount of pain while climbing stairs. 0 being no pain at all and 100 the worst pain possible.
Stair climbing: confidence level | at baseline and after the end of the supplementation period (4-months)
  Participants' confidence when using the staircase will be evaluated using a numerical rating scale.
  Participants will have to answer to the questions:
  Before starting the stair climbing trials: How confident are you that you can go up and down the stairs without falling?
  After the stair climbing trials: Now that you have used the staircase, how confident were you that you would not fall while using it?
  They will answer on a scale from 0 to 10, 0 being not confident at all and 10 being completely confident.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O'Brien, PhD, Study Director — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University - Tom Reilly Building, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No